CLINICAL TRIAL: NCT06888401
Title: Clinico-demographic Profile of the Patient With Pancreaticobiliary Malignancy Undergoing ERCP in a Tertiary Care Center of Nepal: A Cross-sectional Study
Brief Title: Clinico-demographic Profile of the Patient With Pancreaticobiliary Malignancy Undergoing ERCP in a Tertiary Care Center of Nepal
Status: Completed | Type: Observational
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Prakash Sapkota, Principal Investigator, Kathmandu University School of Medical Sciences
Other Study IDs: KUSMS-IRC (39/23)
Record Dates: First submitted 2025-03-11; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cholangiocarcinoma; Bile Duct Carcinoma; Endoscopic Retrograde Cholangio-Pancreatography; Pancreatic Neoplasms
Keywords: Bile duct; Cholangiocarcinoma; Endoscopic Retrograde Cholangiopancreatography; Nepal; Pancreatic Neoplasm
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms; Pancreatic Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ERCP

SUMMARY:
Background Pancreaticobiliary malignancy (PBM) is a group of cancers affecting pancreas and bile duct. The diagnosis is often late and with fatal outcomes. Here, investigators study the clinicodemographic profile of the patients with suspected PBM undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP) at a tertiary care center in Nepal.

Material and Methods Retrospectively, a descriptive cross-sectional study was conducted at the endoscopy unit of the Internal medicine department of Dhulikhel Hospital-Kathmandu University Hospital (DH-KUH) from Jan 2017 to Jan 2023. Patients over 18 years of age with suspected PBM with complete medical records who underwent ERCP were included in our study. The descriptive and correlation statistics were done.

ELIGIBILITY:
Inclusion Criteria:

* above 18years of age.
* those with confirmed pancreaticobiliary malignancies, diagnosed through histopathology from ERCP, or Endoscopic Ultrasound (EUS), or Computerized tomography (CT) guided biopsy, and who underwent ERCP
* those with strong suspicions of malignancy confirmed by clinical, CT scan and ERCP findings, and who also underwent ERCP

Exclusion Criteria:

* those with suspected intrahepatic cholangiocarcinoma, who underwent percutaneous transhepatic cholangiography with biliary drainage
* Those with incomplete hospital records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total population sampling was performed from the medical records of patients fulfilling the inclusion criteria. All the eligible cases that were listed in the medical record of Dhulikhel Hospital from January 2017 to January 2023 were obtained manually. The tally considered patients undergoing multiple ERCP procedures as a single case.
Sampling Method: Non-Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Measurement of risk factors in patients with Pancreaticobiliary Malignancy | 6 years from January 2017 to January 2023.
  The risk factors will be assessed on the basis of physiological parameters like age, dietary habits, smoking and alcohol habits and comorbities.
Measurement of clinical patterns in patients with Pancreaticobiliary Malignancy | 6 years from January 2017 to January 2023.
  The clinical patterns will be assessed on the basis of data collected from self-structured proforma that was used as research tool for data collection based on literature review. The patient information was obtained from hospital records after informed consent.
Measurement of treatment modalities in patients with Pancreaticobiliary Malignancy | 6 years from January 2017 to January 2023.
  The treatment modalities will be assessed with a self-structured proforma which will include the type of treatment modalities like surgical or medical or combined, and the the choice of stent type and technical success of type of stents.

CONTACTS AND LOCATIONS:
Locations (1):
- Kathmandu University School of Medical Sciences, Dhulikhel, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be available upon request from the analysis report.

REFERENCES:
- [Background] Makar M, Zhao E, Tyberg A. Personalized Approach to the Role of Endoscopic Ultrasound in the Diagnosis and Management of Pancreaticobiliary Malignancies. J Pers Med. 2021 Mar 4;11(3):180. doi: 10.3390/jpm11030180. PMID 33806458
- [Background] England RE, Martin DF. Endoscopic and percutaneous intervention in malignant obstructive jaundice. Cardiovasc Intervent Radiol. 1996 Nov-Dec;19(6):381-7. doi: 10.1007/BF02577624. PMID 8994702
- [Background] Mumtaz K, Hamid S, Jafri W. Endoscopic retrograde cholangiopancreaticography with or without stenting in patients with pancreaticobiliary malignancy, prior to surgery. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD006001. doi: 10.1002/14651858.CD006001.pub2. PMID 17636818

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-03-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT06888401/Prot_SAP_ICF_000.pdf